CLINICAL TRIAL: NCT06997185
Title: Communicating Uncertainties Associated With the Benefits and Risks of New Cancer Drugs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Economics and Political Science (Other)
Collaborators: Harvard Medical School / Harvard Pilgrim Health Care Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 540788
Record Dates: First submitted 2025-05-09; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Cancer
Keywords: Cancer; Uncertainty; Prescription drug information
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Single arm trial (Experimental)
  Interventions: Other: Statement communicating uncertainty with a single arm trial
- Limited study duration (long-term benefits and harms) (Experimental)
  Interventions: Other: Statement communicating uncertainty with limited study duration
- Limited study population (generalizability) (Experimental)
  Interventions: Other: Statement communicating uncertainty with a limited study population
- Unvalidated surrogate endpoint (Experimental)
  Interventions: Other: Statement communicating uncertainty with an unvalidated surrogate endpoint
- Treatment effect size (magnitude of benefit) (Experimental)
  Interventions: Other: Statement communicating uncertainty with treatment effect size

INTERVENTIONS:
Other: Statement communicating uncertainty with a single arm trial — Because Zenova has not been compared to other treatments, it is unknown if Zenova is better, the same, or worse than other treatments for non-small cell lung cancer.
  Arms: Single arm trial
Other: Statement communicating uncertainty with limited study duration — Since patients given Zenova were followed for a short time, the longer-term benefits and harms of taking Zenova are unknown.
  Arms: Limited study duration (long-term benefits and harms)
Other: Statement communicating uncertainty with a limited study population — Zenova has not been studied in patients similar to Alex (patients with her race and ethnicity). It is unknown whether Zenova will work and what harms it will have for patients like her.
  Arms: Limited study population (generalizability)
Other: Statement communicating uncertainty with an unvalidated surrogate endpoint — Zenova has only been shown to shrink the size of tumors. It is unknown whether Zenova improves how patients feel or how long they live.
  Arms: Unvalidated surrogate endpoint
Other: Statement communicating uncertainty with treatment effect size — It is unknown whether patients with non-small cell lung cancer will notice an improvement with Zenova.
  Arms: Treatment effect size (magnitude of benefit)

SUMMARY:
This nationally representative randomized survey of US adults will evaluate the effect of using brief statements to communicate different sources of uncertainty about the benefits and harms of new cancer drugs on participants' decisions and understanding.

DETAILED DESCRIPTION:
Many newer cancer drugs are approved before uncertainties with their underlying clinical trial evidence have been adequately studied, in turn making it difficult to accurately determine the drug's benefits and harms. Prescription drug information rarely communicates these uncertainties. In a nationally representative sample of US adults, this study will evaluate the effect of using brief statements to communicate different sources of uncertainty about the benefits and harms of new cancer drugs on participants' decisions and understanding.

In the pre-intervention phase, participants will be given information about a hypothetical new drug approved for the treatment of non-small cell lung cancer. Participants will be asked how likely they would be to take the drug, and how certain they are that the drug will work. Participants will then be randomized to 1 of 5 statements about a source of uncertainty with the drug's evidence that were based on the most common sources of uncertainties with new cancer drugs that are cited in FDA approval decisions: (1) single-arm trial designs, (2) limited study populations (i.e., generalizability of clinical trial evidence), and (3) limited study durations (i.e., long-term benefits and harms). Two additional uncertainties were also included that are frequently mentioned in the scientific literature: (4) the use of unvalidated surrogate endpoints to support new cancer drug approvals, and (5) uncertain treatment effect size (i.e., the magnitude of therapeutic benefit). The post-intervention questions will re-assess participants' decision making and perceptions of uncertainty, as well as their understanding of the uncertainty communicated in the statement.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age and older
* Adults fluent in English
* Adults residing in the United States

Exclusion Criteria:

* Participants who do not meet each of the 3 inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change in decisions | 15-minute survey. Change in decisions is assessed by participants answers to the question pre- and post-intervention.
  "Imagine you were Alex and diagnosed with non-small cell lung cancer. How likely are you to take the new drug, Zenova?"
  4-point Likert scale for decision: very likely; somewhat likely; somewhat unlikely; very unlikely.
Understanding | 15-minute survey. Assessed post-intervention.
  Please answer rate your agreement with the following statements. Zenova works better than other treatments for non-small cell lung cancer Zenova's longer-term benefits and harms are well known Zenova has been studied in patients that are similar to Alex (race and ethnicity) Zenova improves how patients feel or how long they live Zenova has a very large benefit for patients with non-small cell lung cancer
  5-point Likert scale for understanding: strongly disagree; somewhat disagree; neither disagree or agree; somewhat agree; strongly agree.

SECONDARY OUTCOMES:
Change in perception of uncertainty | 15-minute survey. Change in perception of uncertainties is assessed by participants answers to the question pre- and post-intervention.
  "How certain are you that Zenova will work for Alex?"
  4-point Likert scale for perception of uncertainty: very uncertain; somewhat uncertain; somewhat certain; very certain.

OTHER OUTCOMES:
Perceived importance of knowing about uncertainty | 15-minute survey. Assessed post-intervention.
  Was the additional information about Zenova helpful to your decision? 4-point Likert scale: strongly disagree; somewhat disagree; somewhat agree; strongly agree.
  Do you think that uncertainties about drug benefits and harms should always be communicated? 4-point Likert scale: strongly disagree; somewhat disagree; somewhat agree; strongly agree.
  Which of these uncertainties do you think are important to know when deciding about taking a new drug?
  * Unknown whether the drug is better or worse than other treatments.
  * Unknown what the long-term benefits and harms of the drug are.
  * Unknown how well the drug will work for you (for example, someone of your age, of your race, or with your health conditions).
  * Unknown whether the drug will help you feel better or live longer.
  * Unknown whether the drug will make a noticeable difference (the benefits are too small to notice).
    4-point Likert scale: not at all important; somewhat unimportant; somewhat important; very important.

CONTACTS AND LOCATIONS:
Locations (1):
- Harvard Medical School and Harvard Pilgrim Health Care Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-05-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT06997185/Prot_SAP_ICF_000.pdf